CLINICAL TRIAL: NCT06766552
Title: A Multicenter Registry Study Assessing Patient Reported Outcome, Dosing Patterns, and Safety of Vunakizumab in Patients With General Rheumatic Diseases.
Brief Title: A Registry Study Assessing PRO, Dosing Patterns, and Safety of Vunakizumab in Patients With General Rheumatic Diseases.
Acronym: V-MIRACLE
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: z220241396
Record Dates: First submitted 2024-12-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Ankylosing Spondylitis (AS); Psoriatic Arthritis (PsA); Nr-axSpA; Polymyalgia Rheumatica (PMR); Takayasu Arteritis (TAK); Giant Cell Arteritis (GCA); Behcet's Disease; Enthesitis-related Arthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic; Non-Radiographic Axial Spondyloarthritis; Polymyalgia Rheumatica; Takayasu Arteritis; Giant Cell Arteritis; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ankylosing spondylitis, radiographically negative axial spondyloarthritis, psoriatic arthritis, polymyalgia rheumatica, Takayasu arteritis, giant cell arteritis, non-ocular Behcet's disease, and enthesitis-related arthritis are common diseases in rheumatology. Traditional anti-rheumatic drugs are less effective and have greater side effects than biological agents. At present, there has been no large-scale registration study on rheumatic autoimmune diseases such as spondyloarthritis in China. However, data such as patient characteristics, medication patterns, and patient outcome reports of different rheumatology diseases can often serve as a reference for rheumatology clinicians to reasonably select treatment methods for different patients. Therefore, a large-scale registration study is needed to fill the gap in multi-disease registration studies in rheumatology departments in China.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with rheumatic autoimmune diseases such as ankylosing spondylitis/radiologically negative axial spondyloarthritis/psoriatic arthritis/polymyalgia rheumatica/Takayasu arteritis/giant cell arteritis/ non-ocular Behcet's disease/ enthesitis-related arthritis;
2. Currently receiving or planning to receive fulvezinib treatment;
3. Can follow up according to the doctor's advice;
4. Able to understand and sign the informed consent form, understand the purpose of this study, and voluntarily participate in this study.

Exclusion Criteria:

1.Investigator believes will prevent the subject from following and completing the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have been diagnosed with rheumatic autoimmune diseases such as ankylosing spondylitis, radiologically negative axial spondyloarthritis, psoriatic arthritis, polymyalgia rheumatica, Takayasu arteritis, giant cell arteritis, non-ocular Behcet's disease, and enthesitis-related arthritis;
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
European Quality of Life-5 Dimensions Questionnaire （EQ5D） score | From enrollment to the end of treatment at 12 months
  European Quality of Life-5 Dimensions Questionnaire （EQ5D） score： The EQ-5D describes five dimensions: mobility, Self-Care, Usual Activities, Pain/comfort, and Anxiety/Depression, each of which contains five levels: No difficulty, a little difficulty, moderate difficulty, serious difficulty, unable to proceed/with very serious difficulty. Using a utility-value conversion table, the EQ-5D index score can be further calculated.
Pain VAS score | From enrollment to the end of treatment at 12 months
  Pain VAS score (if applicable)：Visual Analogue Scale, The VAS score is indicated by a 10-cm-long straight line, with one end of the line indicating "no pain" (score 0) and the other end indicating "most severe pain" (score 10). Patients marked positions on this line that corresponded to their pain level, and pain was assessed by measuring the distance from the "painless" end to the marked point.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, China